CLINICAL TRIAL: NCT03395444
Title: Double Blind Placebo-controlled Clinical Trial to Assess Pulsed Shortwave Therapy as an Adjunct Pain Therapy & Knee Recovery for Total Knee Arthroplasty
Brief Title: Pulsed Shortwave Therapy Adjunct Pain and Recovery in Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Biel-TKA-001
Record Dates: First submitted 2017-12-21; First posted 2018-01-10 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-12

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): Pulsed shortwave therapy device used as an adjunct therapy immediately on the completion of the operation
  Interventions: Device: pulsed shortwave therapy
- Control Group (Sham Comparator): Sham pulsed shortwave therapy device used as an adjunct therapy immediately on the completion of the operation
  Interventions: Device: pulsed shortwave therapy

INTERVENTIONS:
Device: pulsed shortwave therapy — Pulsed shortwave therapy us the RecoveryRx device. Emits a pulsed signal a the 27.12Mhz wavelength
  Other Names: RecoveryRx

SUMMARY:
This clinical study is designed to assesses the benefit of adding pulsed shortwave therapy to the postoperative pain and recovery protocol following total knee replacement. Pulsed shortwave therapy is a safe adjunct pain therapy for acute and chronic pain.

DETAILED DESCRIPTION:
Despite the recent advances in the understanding of pain mechanisms and the introduction of new drugs and new techniques in the postoperative management, pain after total knee arthroplasty (TKA) is still an unresolved issue. It affects the quality of life and rehabilitation of an important percentage of patients undergoing TKA. A recent study looked at the percentage of patients with chronic knee pain after knee replacement at a minimum of one year following surgery in 272 patients, 107 patients (nearly 40%) reported that they still had persistent pain at one-plus year following surgery. Central sensitization is now well established as an integral factor in many chronic pain states, including the commonly occurring knee and back pain. Many patients undergoing TKA are likely to have a significant degree of Central Sensitization, therefore the likely hood of high pain levels postoperative and persistent long standing pain after TKA is increased in this patient population.

Pulsed shortwave therapy negates central sensitization by imputing new

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for knee osteoarthritis;
* Planned spinal anesthesia; American Society of Anesthesiologists (ASA) physical status I-II;
* Scheduled for unilateral TKA;
* Patients aged 50 to 80 years old.
* Willingness to give written informed consent and willingness to participate in and comply with the study.

Exclusion Criteria:

* Unwillingness of the patient;
* Presence of neuropathic pain or sensory disorders in the leg to be operated on;
* Intolerance to the study drugs;
* Failure of spinal anesthesia;
* Previous major knee surgery, re-operation or trauma to the knee within the study period.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogue Pain | Change in pain levels over 3 months
  The visual analog scale (VAS) has been used extensively for rating pain intensity in previous studies. Postoperative pain at 2, 6, 10, 18, 26, 34, 42, 50, 58, 64, and 72 hours after surgery will be recorded using a 10-cm horizontal line with 1-cm vertical lines at each end labeled "no pain" (left side) and "worst possible pain" (right side). VAS scores will also be recorded also at day 4, 7, 14 and 28 and finally at three months. Different time point assessments are being conducted to look at the change in pain level from baseline through recovery.

SECONDARY OUTCOMES:
The Oxford Knee Score | 3 months
  The Oxford Knee Score (OKS) is a 12-item patient-reported PRO specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is short, reproducible, valid and sensitive to clinically important changes.
The Knee Injury and Osteoarthritis Outcome Score | 3 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
Pain Pressure Threshold | 3 months
  Pain Pressure Threshold, is used routinely in clinical practice to assess pain sensitivity from musculoskeletal pain to indicate the level of pain sensitivity in individuals to central sensitization of the nervous system. Testing will occur locally above the effected knee as well as peripherally on the distal interphalangeal joint.
The Pain and Sleep Questionnaire three-item index | 3 months
  The Pain and Sleep Questionnaire three-item index (PSQ-3): A reliable and valid measure of the impact of pain on sleep in chronic nonmalignant pain of various etiologies.
Active Range of Motion | 3 months
  Active range of motion (A-ROM) is an important component of the assessment of total knee replacement (TKR) outcome. The goal of knee replacement recovery is to achieve flexion of 135 degrees. Range of motion will be measured by observational method by two separate individuals.
Analgesic medication use | 28 days
  Analgesic medication use for the postoperative period of 7 days as well as a further 21 days will be recorded - 28 day total.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Tabbouche, Pharm D, Study Director — New Mazloum Hospital; Raed El Hassan, Dr, Principal Investigator — New Mazloum Hospital
Locations (1):
- New Mazloum Hospital, Tripoli, Lebanon

IPD SHARING:
Plan to Share IPD: No